CLINICAL TRIAL: NCT00408785
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of BOTOX? (Botulinum Toxin Type A) in Subjects With Glabellar Lines
Brief Title: A Study Of BOTOX For The Treatment Of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107457
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2011-11

CONDITIONS: Glabellar Lines
Keywords: Botulinum Toxin Type A; safety; efficacy; glabellar lines
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Injection
  Interventions: Drug: Botulinum Toxin Type A
- B (Placebo Comparator): Injection
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Botulinum Toxin Type A — botulinum toxin type A 100 units, human serum albumin 0.5 mg, sodium chloride 0.9 mg
  Arms: A
Drug: sodium chloride — sodium chloride 0.9 mg
  Arms: B

SUMMARY:
This is a Multicenter, double-blind, randomized, placebo-controlled, parallel-group comparative study to confirm the efficacy and safety of BOTOX 20 units single injection for the Chinese patients with glabellar lines. The subjects will receive a single intramuscular treatment consisting of 5 injections of either BOTOX? 20U or placebo.

ELIGIBILITY:
Inclusion criteria:

* Male and female adult with Glabellar lines of at least moderate severity at maximum frown by investigator's assessment.

Exclusion criteria:

* Patients with systemic nerve conduction junction disorder or patients with infection or other skin disease/surgery at injection sites will not be eligible.
* Patient with severe complications related to heart, kidney, liver disease or respiratory system will not be eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256
Dates: Start 2006-11-01 (Actual); Primary Completion 2007-05-09 (Actual); Study Completion 2007-05-09 (Actual)

PRIMARY OUTCOMES:
The investigator's rating of Glabellar line severity at maximum frown | Day 30 after injection

SECONDARY OUTCOMES:
Investigator's rating of Glabellar line severity at rest, subject's global assessment of change in appearance of glabellar lines, the subject's perception of age and safety evaluations. | Day 7, 30, 60, 90, 120 after injection

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- China (2):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai